CLINICAL TRIAL: NCT00276302
Title: A Phase 1, Safety Assessment and Pharmacokinetic Study of IPI-504 in Patients With Either Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GIST) or Advanced or Metastatic Soft Tissue Sarcomas (STS)
Brief Title: Safety Study of IPI-504 in Patients With Gastrointestinal Stromal Tumors (GIST) or Soft Tissue Sarcomas (STS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Krista McKee, MEd, MPH, Infinity Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-02
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Gastrointestinal Stromal Tumors; Soft Tissue Sarcomas
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Schedule A: Doses occur on Days 1, 4, 8, and 11 followed by 10 days with no study drug administration.
  Interventions: Drug: IPI-504
- 2 (Experimental): Schedule B: Doses occur on Days 1, 4, 8, 11, 15, and 18 (twice weekly for 3 weeks continuously).
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — IV administration of IPI-504 for 21-day cycles. Two different schedules of treatment will be tested. On Schedule A, doses occur on Days 1, 4, 8, and 11 followed by 10 days with no study drug administration. On Schedule B, doses occur on Days 1, 4, 8, 11, 15, and 18, or twice weekly for 3 weeks continuously.
  For both Schedule A and B doses will be administered ≥ 72 hours apart.

SUMMARY:
The primary objectives of the study are:

* Determine the safety and maximum tolerated dose (MTD) of IPI-504 in GIST and STS patients who have failed prior therapies
* Recommend a dose for subsequent studies of IPI-504

DETAILED DESCRIPTION:
IPI-504 is a novel, water-soluble analog of 17-AAG and a potent inhibitor of Hsp90. Hsp90's role in the cell is to control the proper folding, function, and viability of various "client" proteins. Many of these client proteins (such as AKT, Her-2, Bcr-Abl, PDGFR-α, and c-Kit) are oncoproteins or important cell signaling proteins. In patients with GIST, mutations in the tyrosine kinase receptor Kit play a critical role in the pathogenesis of this disease. Inhibition of Kit signaling with the tyrosine kinase inhibitor Imatinib (IM) is a very effective treatment for GIST patients. However, new mutations arise in Kit conferring resistance to IM treatment which results in disease progression. Kit is a client protein of Hsp90 and is sensitive to IPI-504. In Soft Tissue Sarcomas, there may be genetic abnormalities that lead to the expression of certain proteins that drive the growth of cancer. These cancer-driving proteins may be stimulated by HSP90. This provides a scientific rationale for Phase 1 clinical testing of IPI-504 in patients with advanced GIST and STS who have failed prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of GIST or STS
* Failed prior therapies
* ECOG performance status of 0-2
* Ability to adhere to the study visit schedule and all protocol requirements

Exclusion Criteria:

* Previous treatment with 17-AAG, DMAG, or other known Hsp90 inhibitor
* Participation in any investigational drug study or treatment with any other kinase inhibitor therapy within 2 weeks preceding start of treatment
* Concurrent radiation therapy is not permitted
* Concurrent treatment with any agent that alters CYP3A activity
* Concurrent treatment with any agent that may prolong the QTc interval
* Myocardial infarction or active ischemic heart disease within 6 months
* History of arrhythmia
* Baseline QTc >450
* Grade 3 or greater peripheral neuropathy
* Renal insufficiency, serum creatinine >1.5 x ULN
* Platelets < 100,000 mm3
* AST and / or ALT > 2.5 x ULN
* ANC <1,500 cells/mm3
* Alkaline phosphatase > 2.5 x ULN
* Amylase and lipase > 1.5 x ULN
* Hemoglobin < 9.0 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and maximum tolerated dose (MTD) of IPI-504 in GIST and STS patients who have failed prior therapies | 18 months
To recommend a dose for subsequent studies of IPI-504 | 18 months

SECONDARY OUTCOMES:
To examine the pharmacokinetic (PK) parameters of IPI-504 in GIST and STS patients | 18 months
To assess in a preliminary way the potential anti-tumor activity of IPI-504 in GIST and STS. | 18 months
To explore potential pharmacodynamic (PD) markers of biologic activity of IPI-504 in GIST and STS. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: George D Demetri, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (4):
  - Premiere Oncology, Scottsdale, Arizona
  - Premiere Oncology, Santa Monica, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hosptials, Ann Arbor, Michigan
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- See also: Gist Support International — http://www.gistsupport.org/
- See also: Life Raft Group — http://www.liferaftgroup.org/